CLINICAL TRIAL: NCT06790628
Title: Assessment of Facial Symmetry Following Fibula Free Flap Fixated in a Prosthetically Favorable Position Versus the Inferior Border Position for Mandibular Reconstruction: a Randomized Controlled Trial.
Brief Title: Assessment of Facial Symmetry Following Fibula Free Flap Fixated in a Prosthetically Favorable Position Versus the Inferior Border Position for Mandibular Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Ahmed Sakr, Ph.D. Candidate in Oral & Maxillofacial surgery departement., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OMFS 3-3-60
Record Dates: First submitted 2025-01-17; First posted 2025-01-24 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Mandible Reconstruction
Keywords: Segmental mandibular defect; mandibular reconstruction; fibula free flap; dental implants; facial symmetry; face scan.

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mandibular reconstruction with fibula free flap fixated in inferior border level. (Active Comparator): Fixation of the fibula in the inferior border level (conventional position).
  Interventions: Procedure: Fibula free flap
- Mandibular reconstruction with fibula free flap fixated in the alveolar level. (Active Comparator): Fixation of the fibula in the alveolar level (prosthetically favorable position) leaving 15-17mm till the opposing teeth.
  Interventions: Procedure: Fibula free flap

INTERVENTIONS:
Procedure: Fibula free flap — surgical technique used in reconstructive surgery where a segment of the fibula bone, along with its blood vessels, is taken from the lower leg and transplanted to reconstruct defects in the mandible due to its length, strength, and ability to support dental implants.
  The blood vessels are connected to nearby vessels at the reconstruction site to ensure the bone's survival and integration.
  The procedure is highly versatile and often referred to as the "gold standard" for mandibular reconstruction.

SUMMARY:
The study aims to evaluate facial symmetry outcomes after mandibular reconstruction using fibula free flaps, comparing two fixation techniques: the prosthetically favorable position (alveolar level) and the conventional position (inferior border level).

DETAILED DESCRIPTION:
The study aims to evaluate facial symmetry outcomes after mandibular reconstruction using fibula free flaps, comparing two fixation techniques: the prosthetically favorable position (alveolar level) and the conventional position (inferior border level).

Design:

A randomized controlled trial with parallel groups and a 1:1 allocation ratio. The study will assess facial symmetry and patient satisfaction over 12 months post-surgery.

Population:

Patients requiring mandibular reconstruction due to conditions like tumors, trauma, or osteomyelitis, with mandibular defects greater than 9 cm.

Interventions:

Group 1: Fibula free flap fixated at the alveolar level (prosthetically favorable position).

Group 2: Fibula free flap fixated at the inferior border level (conventional position).

Setting:

Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Cairo University.

Duration:

Follow-up over 12 months post-surgery, with key data collection points at baseline, 3 days, 1 week, 1 month, 6 months, and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patient who requires mandibular resection due to tumor, trauma, osteomyelitis or osteoradionecrosis.
* Patient with Mandibular defect >9 cm.

Exclusion Criteria:

- Patients with systemic condition counteracting with the surgical procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Facial Symmetry | 6-12 months
  Tool: 3D Stereophotogrammetry face scan. Unit: RMSD: root mean square deviation (Millimeters). Method: superimposition of the face scan color maps on Materialise's Interactive Medical Image Control System (MIMICS) Software.

SECONDARY OUTCOMES:
Patient Satisfaction. | 6-12 months
  Tool: Questionnare (Visual analogue scale) Unit: Scale (1-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Oral & Maxillofacial department - Faculty of Dentistry - Cairo University., Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided